CLINICAL TRIAL: NCT05218265
Title: Criteria and Potential Predictors of Severity in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmad Abbas, Assistant professor of chest diseases, Zagazig University
Other Study IDs: 9229
Record Dates: First submitted 2022-01-30; First posted 2022-02-01 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: routine laboratory tests — Complete blood count (CBC), coagulation profile, serum biochemical tests (including renal and liver function, and electrolytes), laboratory investigation to assess severity of COVID-19: lactate dehydrogenase (LDH), myocardial enzymes (CPK-MB), serum ferritin, D dimer and arterial blood gases analysis

SUMMARY:
This is an observational cross sectional study included 202 patients diagnosed to have COVID-19. The study was conducted at Zagazig University Isolation Hospitals from the period of March 2020 to June 2021. The study was approved by Zagazig University Ethics Committee (number 9229). A written informed consent was obtained from all participants.

Inclusion criteria:

The study includes laboratory confirmed COVID-19 patients (confirmed by real-time polymerase chain reaction) admitted l during the period of the study.

The patients were classified into two groups, group A included mild/moderate cases, group B included severe/critical cases according to the following criteria.

Severity of COVID-19 was graded as follows: mild; mild clinical symptoms, no pneumonia on lung CT; moderate: fever, cough and lung CT with pneumonia; severe: respiratory distress (respiratory rate > 30 /min, oxygen saturation (O2Sat) ≤ 93 percent at rest and/or ratio of arterial oxygen partial pressure to fractional inspired oxygen ≤300 mmHg (PaO2/FIO2); and critical: aforementioned criteria of respiratory failure receiving mechanical ventilation, shock, and/or organ failure other than lung and/or intensive care unit (ICU) hospitalization.

All participants were subjected to full history taking including smoking history and comorbidity profile. Clinical symptoms including: fever, cough, dyspnea, myalgia, hemoptysis, sore throat, diarrhea, loss of smell and anorexia were recorded. Radiological assessment by initial chest x ray then CT chest as possible and appropriate. Routine laboratory investigations: Complete blood count (CBC), coagulation profile, serum biochemical tests (including renal and liver function, and electrolytes), laboratory investigation to assess severity of COVID-19: lactate dehydrogenase (LDH), myocardial enzymes (CPK-MB), serum ferritin, D dimer and arterial blood gases analysis. Patients were followed up for the need for ICU and mechanical ventilation (MV), duration till conversion, total length of stay and final outcome whether survived or died were recorded.

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed COVID-19 patients (confirmed by real-time polymerase chain reaction) admitted during the period of the study.

Exclusion Criteria:

* age less than 18
* refusal to participate
* referral to other hospital within 24 hours of admission
* missing data registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational cross sectional study included 202 patients diagnosed to have COVID-19. The study was conducted at Zagazig University Isolation Hospitals from the period of March 2020 to June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
assessing severity of COVID-19 | 30 days from admission
  Severity of COVID-19 was graded as follows: (1) mild; mild clinical symptoms, no pneumonia on lung CT; (2) moderate: fever, cough and lung CT with pneumonia; (3) severe: respiratory distress (respiratory rate > 30 /min, oxygen saturation (O2Sat) ≤ 93 percent at rest and/or ratio of arterial oxygen partial pressure to fractional inspired oxygen ≤300 mmHg (PaO2/FIO2); and (4) critical: aforementioned criteria of respiratory failure receiving mechanical ventilation, shock, and/or organ failure other than lung and/or intensive care unit (ICU) hospitalization [according to 16.National Health Commission of China. The novel coronavirus pneumonia diagnosis and treatment program, 7th version. China. 2020.http://www.nhc.gov.cn/yzygj/s7653p/202003/46c9294a7dfe4cef80dc7f5912eb1989.shtml. Accesed 04 Apr.]

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of medicine Chest Department, Zagazig, Asharqia, Egypt